CLINICAL TRIAL: NCT07114523
Title: Effect of Collagen Membranes on Distal Periodontal Healing of Second Molars After Impacted Mandibular Third Molar Surgery: A Randomized Controlled Trial
Brief Title: Effect of Collagen Membranes on Distal Periodontal Healing of Second Molars After Impacted Mandibular Third Molar Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Lam Cu Phong, lecturer, clinical professor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3566/DHYD-HDDD
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Defect

STUDY DESIGN:
Intervention Model Description: This type of interventional study in dentistry is referred to as a split-mouth design. In this design, the intervention subjects have bilaterally symmetrical conditions within the oral cavity, allowing one side to serve as the intervention group while the contralateral side serves as the control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): apply collagen membrane on distal surface of second molar after third molar surgery
  Interventions: Procedure: collagen membrane
- control (Active Comparator): standard third molar surgery without any application
  Interventions: Procedure: third molar surgery

INTERVENTIONS:
Procedure: collagen membrane — collagen membrane apply to distal surface of second molar after third molar surgery
  Arms: study
Procedure: third molar surgery — standard third molar surgery without any additional application
  Arms: control

SUMMARY:
Impacted mandibular third molars can cause various complications to the adjacent second molars, such as dental caries, periodontitis, or root resorption. These complications often progress silently and asymptomatically. A typical scenario involves a mesioangularly impacted third molar exerting pressure on the distal alveolar bone of the second molar, resulting in persistent food impaction that is difficult for patients to clean. Furthermore, the surgical removal of deeply impacted or severely angulated mandibular third molars often requires bone removal in the area adjacent to the second molar. These factors may exacerbate distal periodontal defects of the second molar, especially in individuals over the age of 25. This research focuses on evaluating the effectiveness of a new-generation collagen membrane in promoting healing after the extraction of impacted mandibular third molars in patients at risk of distal periodontal tissue damage to the second molars

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25 years or older.
* Patients with mesioangular or horizontally impacted mandibular third molars. The highest point of mandibular third molars are lower than the occlusal surface of adjacent second molars (classified B, C according to Pell - Gregory's category).
* Patients with symmetrical lower third molars on both sides with same classification according to Pell - Gregory's category. The difference of third molars inclination on both side is not more than 15°.
* Patients with lower second molars on both sides have no cavities or fillings that affect the determination of the cemento-enamel junction.
* Patients are explained, counseled clearly and sign their consent to participate in the study.

Exclusion Criteria:

* Patients with coagulation or immune disorders.
* Patients allergic to local anesthetics (Lidocaine 2% with Adrenaline 1:100,000) or any drugs used in the study.
* Patients allergic to products or food derived from pigs.
* Pregnant or breastfeeding patients.
* Patients who smoke.
* Patients with systemic conditions that contraindicate surgical procedures.
* Patients with clinical or radiographic signs suggestive of tumors (benign or malignant) associated with or in proximity to the mandibular third molar.
* Patients with missing mandibular second molars.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Distal periodontal tissue status | preoperative (T0), 3rd moth after surgery (T3) and 6th month after surgery (T6)
  distal periodontal tissue status was assessed using variables of pocket depth

SECONDARY OUTCOMES:
Distal bone level | at the time of the end of surgery (T0'), 3rd month after surgery (T3), and 6th month after surgery (T6).
  The variable was determined by measuring the distance from the CEJ of mandibular second molar to the highest point of the alveolar crest, performed with the periapical radiograph using the parallel technique, standardized with a film holder and a stent with a 5 mm steel segment

OTHER OUTCOMES:
Postoperative pain | on the 1st, 3rd, 7th day after surgery
  Postoperative pain was assessed by patient using the VAS (Visual Analog Scale) on the 1st, 3rd, 7th day after surgery. The VAS pain assessment scale is a 100 mm long line with 2 endpoints defined as "no pain" on the left side and "maximum pain" on the right side. The patient will record his/her pain level by marking a point on the line, the pain point will be the distance measured from the left endpoint to the point marked by patient.
Postoperative swelling | on the 1st, 3rd, 7th day after surgery
  Facial swelling was assessed by the patient using the modified VAS scale of Pasqualini et al (2005) on the 1st, 3rd, 7th day after surgery. The scale consisted of 6 levels from 0 (no swelling) to 5 (severe swelling), patient will choose the corresponding level of swelling.
Soft tissue healing | on the 7th day after surgery
  Soft tissue healing was assessed using Healing index of Landry, Turnbull, and Howley on the 7th day after surgery. The scale consists of 5 grades, from grade 1 (very poor healing) to grade 5 (excellent healing) based on signs of tissue color, bleeding, presence of granulation tissue, presence of pus, and degree of epithelialization.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol